CLINICAL TRIAL: NCT00337610
Title: A Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Efficacy of the Addition of Sitagliptin to Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Therapy
Brief Title: Sitagliptin Metformin Add-on Study in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-053; 2006_017
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Results first posted 2010-05-27 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- sitagliptin 100 mg once a day (q.d.)/metformin ≥1500 mg a day (Experimental)
  Interventions: Drug: sitagliptin 100 mg q.d./metformin ≥ 1500 mg/day
- sitagliptin 100 mg placebo q.d./ metformin ≥ 1500 mg/day (Placebo Comparator)
  Interventions: Drug: comparator: placebo to match sitagliptin 100 mg q.d./metformin ≥ 1500 mg/day

INTERVENTIONS:
Drug: sitagliptin 100 mg q.d./metformin ≥ 1500 mg/day — Patients will receive blinded sitagliptin 100 mg q.d. and open-label metformin ≥ 1500 mg/day for up to 30 weeks. Sitagliptin 100 mg q.d. and metformin ≥ 1500 mg/day will be administered as oral tablets.
  Other Names: Januvia
  Arms: sitagliptin 100 mg once a day (q.d.)/metformin ≥1500 mg a day
Drug: comparator: placebo to match sitagliptin 100 mg q.d./metformin ≥ 1500 mg/day — Patients will receive placebo to match sitagliptin 100 mg q.d. and open-label metformin ≥ 1500 mg/day for up to 30 weeks. Sitagliptin 100 mg q.d. and metformin ≥ 1500 mg/day will be administered as oral tablets.
  Arms: sitagliptin 100 mg placebo q.d./ metformin ≥ 1500 mg/day

SUMMARY:
A clinical study to determine the safety and efficacy of sitagliptin in patients with Type 2 Diabetes Mellitus who have inadequate glycemic (blood sugar) control on metformin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has type 2 diabetes mellitus
* Males
* Females who are highly unlikely to become pregnant
* Patients poorly controlled while taking one or two oral antidiabetic medications

Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or history of ketoacidosis
* Patient required insulin therapy within the prior 8 weeks
* Patient is on or has been taking Thiazolidinediones (TZDs) such as Actos® (pioglitazone) or Avandia® (rosiglitazone) or is on or has been taking Byetta® (exenatide) within the prior 12 weeks of the screening visit

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Raz I, Chen Y, Wu M, Hussain S, Kaufman KD, Amatruda JM, Langdon RB, Stein PP, Alba M. Efficacy and safety of sitagliptin added to ongoing metformin therapy in patients with type 2 diabetes. Curr Med Res Opin. 2008 Feb;24(2):537-50. doi: 10.1185/030079908x260925. PMID 18194595

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 21-Aug-2006; Last Patient Last Visit: 15-Aug-2007; Twenty-four medical clinics worldwide (12 in the United States, 2 in Israel, 3 in Mexico, 3 in Peru, and 4 in Austria).
Pre-assignment Details: Patients 18-78 years on oral single antihyperglycemic agent (AHA) (hemoglobin A1C [A1C] ≥8%) or metformin-based dual combination therapy (A1C 7.5-10.5%) were eligible to participate. Eligible patients underwent an up to 12-week metformin dose-titration/dose-stable period followed by a 2-week placebo run-in period prior to randomization.
Groups:
- Sitagliptin 100 mg: The Sitagliptin 100 mg group includes data from patients randomized to receive treatment with 100 mg oral tablets of sitagliptin once daily in addition to ongoing treatment with open-label metformin ≥ 1500 mg/day.
- Placebo: The Placebo group includes data from patients randomized to receive treatment with oral tablets of sitagliptin-matching placebo once daily in addition to ongoing treatment with open-label metformin ≥ 1500 mg/day.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg | Placebo
Started | 96 | 94
Completed Week 18 | 89 | 82
Completed | 79 | 80
Not Completed | 17 | 14
Not completed — Adverse Event | 2 | 2
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 6 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Placebo | Total
Number analyzed (Participants) | 96 | 94 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (9.5) | 56.1 (9.5) | 54.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 55 | 102
  Male | 49 | 39 | 88
Race/Ethnicity, Customized [Number; unit: participants]
  White | 40 | 44 | 84
  Black | 3 | 1 | 4
  Hispanic | 31 | 24 | 55
  Asian | 1 | 0 | 1
  Other | 21 | 25 | 46
2-Hour Post-Meal Glucose (2 hr PMG) [Mean (Standard Deviation); unit: mg/dL] | 288.7 (74.8) | 286.7 (61.7) | 287.7 (68.5)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 201.1 (46.2) | 198.2 (44.6) | 199.7 (45.3)
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent] | 9.3 (0.9) | 9.1 (0.8) | 9.2 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 18
Description: A1C was measured as a percent. Thus, this change from baseline reflects the Week 18 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 18
Population: The full-analysis-set (FAS) population included all patients with at least one dose of double-blind study therapy, and with a baseline value and ≥1 postbaseline value for this outcome. Data following glycemic rescue were treated as missing. Missing data were handled using the last observation carrying forward (LOCF) method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 95 | 92
Percent | -1.00 [-1.24 to -0.75] | 0.02 [-0.23 to 0.27]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; prior anti-hyperglycemic agent (AHA) [medication] (on Monotherapy AHA or on Metformin-based combination therapy); Mean Difference (Net) = -1.02, 95% CI [-1.36 to -0.67], Standard Deviation 1.19

2. Secondary Outcome: Change From Baseline in FPG at Week 18
Description: Change from baseline at Week 18 is defined as Week 18 FPG minus Week 0 FPG.
Time Frame: Baseline and Week 18
Population: The full-analysis-set (FAS) population included all patients with at least one dose of double-blind study therapy, and with a baseline value and ≥1 postbaseline value for this outcome. Data following glycemic rescue were treated as missing. Missing data were handled using the LOCF method.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 96 | 92
mg/dL | -32.0 [-40.6 to -23.3] | -6.5 [-15.1 to 2.2]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; prior anti-hyperglycemic medication (on Monotherapy AHA or on Metformin-based combination therapy); Mean Difference (Net) = -25.5, 95% CI [-37.7 to -13.3], Standard Deviation 42.2

3. Secondary Outcome: Change From Baseline in 2 Hr-PMG at Week 18
Description: Change from baseline at Week 18 is defined as Week 18 minus Week 0.
Time Frame: Baseline and Week 18
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 79 | 74
mg/dL | -67.6 [-82.1 to -53.2] | -13.5 [-28.2 to 1.2]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -54.1, 95% CI [-74.7 to -33.6], Standard Deviation 63.8

4. Secondary Outcome: Change From Baseline in A1C at Week 30
Description: A1C was measured as a percent. Thus, this change from baseline reflects the Week 30 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 30
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 95 | 92
Percent | -0.98 [-1.25 to -0.70] | 0.04 [-0.24 to 0.31]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.01, 95% CI [-1.40 to -0.62], Standard Deviation 1.34

ADVERSE EVENTS:
Time Frame: Weeks 0 to 30
Arm/Group | Sitagliptin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/96 | 5/94
Other Adverse Events (participants affected / at risk) | 18/96 | 29/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=96) | Placebo (N=94)
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=96) | Placebo (N=94)
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Nasopharyngitis (Infections and infestations) | 7 | 6
Pharyngitis (Infections and infestations) | 4 | 6
Blood Glucose Increased (Investigations) | 6 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.